CLINICAL TRIAL: NCT00342134
Title: Immunological Mechanisms of Immune Ablation and Autologous Hematopoietic Stem Cell Transplantation in Secondary Progressive Multiple Sclerosis
Brief Title: Immunological Mechanisms of Hematopoietic Stem Cell Transplantation in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999902196; 02-N-N196
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-04

CONDITIONS: Multiple Sclerosis
Keywords: Demyelination; Inflammation; Immunosuppression; Autoimmunity; Bone Marrow; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Inflammation; Autoimmune Diseases

INTERVENTIONS:
Procedure: Stem Cell Transplanataion

SUMMARY:
Our goal is the elucidation of the mechanisms of action of autologous hematopoietic stem cell transplant (HSCT) and immunoablation by high-dose cyclophosphamide in multiple sclerosis (MS).

The molecular pathogenesis of multiple sclerosis is poorly understood although T-cell mediated immune destruction of myelin is thought to be an important element. We hypothesize, and the results of previous studies suggest, that radical immuno-ablation characterized by a profound T cell depletion can arrest the progression of disease. Patients with MS with poor prognosis based on the rate of progression and refractoriness to approved treatments (interferon-beta, glatiramer acetate) will be enrolled in clinical trials at the collaborating institution (NWU-Dr. R. Burt; Dr. D Kerr, JHU) and will receive either immune ablation with cyclophosphamide and the antibody Campath-1 followed by reconstitution with autologous peripheral blood stem cells, a procedure similar to autologous bone marrow transplantation, or high-dose cyclophosphamide treatment without stem cell rescue. While the overall treatment-related mortality worldwide is approximately 10%, the collaborating institution and investigators have an outstanding safety record in performing the procedure with no fatal adverse events after having transplanted more than 30 transplants with a previously more aggressive regimen than the one that is in use now. The underlying rationale for this treatment is that immuno-ablation could eliminate myelin-reactive T cells which, in disease-susceptible individuals, may have been activated by previous exposure to environmental agents or other acquired mechanisms of immune dysregulation.

In the proposed study we plan to address whether HSCT or immunoablation without stem cell rescue act beneficially in MS via the eradication of myelin-reactive T cells and reconstitution of a functional and non-autoimmune immune repertoire. To achieve this goal, we will compare peripheral blood T cell reactivities to myelin antigens before and after the treatment in 34 patients with MS. In parallel, to identify potential disease-mediating cells that do not recognize these myelin antigens, we will search for clonally expanded cells in the blood of MS patients before treatment employing molecular analysis of T cell receptor repertoire. Expanded T cell clones will be tracked during post-transplant follow-up of patients. If the eradication of certain clonotypes resulting from immuno-ablation correlates with disease remission, we will attempt to isolate these cells in culture from pre-treatment samples and determine their specificity using combinatorial peptide libraries. We would use the same approach in case of reappearance or new clonal expansions concomitant to disease relapses. We will combine these studies with a broader, unbiased approach that employs microarray technology to identify potential changes in gene expression profiles. This approach may also lead to the identification of novel therapeutic targets for pharmacological treatment.

DETAILED DESCRIPTION:
Our goal is the elucidation of the mechanisms of action of autologous hematopoietic stem cell transplant (HSCT) and immunoablation by high-dose cyclophosphamide in multiple sclerosis (MS).

The molecular pathogenesis of multiple sclerosis is poorly understood although T-cell mediated immune destruction of myelin is thought to be an important element. We hypothesize, and the results of previous studies suggest, that radical immuno-ablation characterized by a profound T cell depletion can arrest the progression of disease. Patients with MS with poor prognosis based on the rate of progression and refractoriness to approved treatments (interferon-beta, glatiramer acetate) will be enrolled in clinical trials at the collaborating institution (NWU-Dr. R. Burt; Dr. D Kerr, JHU) and will receive either immune ablation with cyclophosphamide and the antibody Campath-1 followed by reconstitution with autologous peripheral blood stem cells, a procedure similar to autologous bone marrow transplantation, or high-dose cyclophosphamide treatment without stem cell rescue. While the overall treatment-related mortality worldwide is approximately 10%, the collaborating institution and investigators have an outstanding safety record in performing the procedure with no fatal adverse events after having transplanted more than 30 transplants with a previously more aggressive regimen than the one that is in use now. The underlying rationale for this treatment is that immuno-ablation could eliminate myelin-reactive T cells which, in disease-susceptible individuals, may have been activated by previous exposure to environmental agents or other acquired mechanisms of immune dysregulation.

In the proposed study we plan to address whether HSCT or immunoablation without stem cell rescue act beneficially in MS via the eradication of myelin-reactive T cells and reconstitution of a functional and non-autoimmune immune repertoire. To achieve this goal, we will compare peripheral blood T cell reactivities to myelin antigens before and after the treatment in 34 patients with MS. In parallel, to identify potential disease-mediating cells that do not recognize these myelin antigens, we will search for clonally expanded cells in the blood of MS patients before treatment employing molecular analysis of T cell receptor repertoire. Expanded T cell clones will be tracked during post-transplant follow-up of patients. If the eradication of certain clonotypes resulting from immuno-ablation correlates with disease remission, we will attempt to isolate these cells in culture from pre-treatment samples and determine their specificity using combinatorial peptide libraries. We would use the same approach in case of reappearance or new clonal expansions concomitant to disease relapses. We will combine these studies with a broader, unbiased approach that employs microarray technology to identify potential changes in gene expression profiles. This approach may also lead to the identification of novel therapeutic targets for pharmacological treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females between the ages of 18 and 70 years, inclusive.

Diagnosis of clinically definite MS according to the McDonald Criteria.

Must have been on conventional immunomodulatory treatment (interferon beta or glatiramer acetate for at least 3 months OR have not tolerated conventional treatment OR have refused to start conventional treatment).

Two or more total gadolinium enhancing lesions on each of two pretreatment MRI scans at screening and enrollment OR one large enhancing lesion measuring at least 1 cm refractory treatment with IV steroids on each of the two pre-treatment scans.

Subject must have EDSS ranging from 1.5 to 6.5.

Subject must have had at least one clinical exacerbation in the last year, and this must have occurred after having been on Avonex, Betaseron, Copaxone or Rebif therapy for at least 3 months. This does not apply if subject has refused to start conventional therapy.

Subject must have had a sustained (greater than or equal to 3 months) increase of greater than or equal to 1.0 on the EDSS (historical estimate allowed) between 1.5 and 5.5 or greater than or equal to 0.5 between 5.5 and 6.5 in the preceding year.

Written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Women of childbearing potential should have a negative pregnancy test prior to entry in to the study.

EXCLUSION CRITERIA:

Any risk of pregnancy - ALL female patients must have an effective means of birth control or be infertile due to hysterectomy, fallopian tube surgery, or premature menopause.

Cardiac ejection fraction of less than 45 percent.

Serum creatinine greater than 2.0.

Patients who are pre-terminal or moribund.

Bilirubin greater than 2.0, transaminases greater than 2 times normal.

Patients with EDSS less than 1.5 or greater than 6.5.

Patients with pacemakers or implants who cannot get serial MRIs.

Patients with active infections until infection is resolved.

Patients with WBC count less than 3000 cells per microliter, platelets less than 100,000 cells per microliter and untransfused hemoglobin less than 10 grams per deciliter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2002-05-01; Primary Completion 2011-05-04 (Actual); Study Completion 2011-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Background] Acha-Orbea H, Mitchell DJ, Timmermann L, Wraith DC, Tausch GS, Waldor MK, Zamvil SS, McDevitt HO, Steinman L. Limited heterogeneity of T cell receptors from lymphocytes mediating autoimmune encephalomyelitis allows specific immune intervention. Cell. 1988 Jul 15;54(2):263-73. doi: 10.1016/0092-8674(88)90558-2. PMID 2455603
- [Background] Bielekova B, Muraro PA, Golestaneh L, Pascal J, McFarland HF, Martin R. Preferential expansion of autoreactive T lymphocytes from the memory T-cell pool by IL-7. J Neuroimmunol. 1999 Dec;100(1-2):115-23. doi: 10.1016/s0165-5728(99)00200-3. PMID 10695722
- [Background] Burns FR, Li XB, Shen N, Offner H, Chou YK, Vandenbark AA, Heber-Katz E. Both rat and mouse T cell receptors specific for the encephalitogenic determinant of myelin basic protein use similar V alpha and V beta chain genes even though the major histocompatibility complex and encephalitogenic determinants being recognized are different. J Exp Med. 1989 Jan 1;169(1):27-39. doi: 10.1084/jem.169.1.27. PMID 2462609